CLINICAL TRIAL: NCT06716268
Title: Dynamics of Pelvic Floor Muscles With Different Phonation Patterns Among Female Students: An Observational Study
Brief Title: Dynamics of Pelvic Floor Muscles With Different Phonation Patterns Among Female Students
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nesma Aziz Abd Elgany, principal investigator, Cairo University
Other Study IDs: P.T.REC/012/005285
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Pelvic Floor Dyssynergia; Phonation Disorder
MeSH Terms: conditions — Dysphonia | interventions — Phonation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Twenty healthy female university students: They will be selected from the faculty of physical therapy ,Cairo university
  Interventions: Other: phonation and respiratory tasks

INTERVENTIONS:
Other: phonation and respiratory tasks — Participants performed various tasks to evaluate pelvic floor muscle activity and displacement. These included a maximum voluntary contraction ("cutting off the flow of urine mid-stream"), a pelvic floor strain ("bearing down for a bowel movement"), and the Valsalva maneuver to clear the Eustachian tubes. Additionally, phonation and respiratory exercises were conducted, such as producing the "ah" sound at different pitches, open-mouth exhalation, coughing, and semi-occluded vocal tract (SOVT) exercises using a small coffee straw, commonly used in singing warm-ups to enhance vocal efficiency. Each task lasted 3 seconds, with 1-minute rest intervals to assess their impact on pelvic floor displacement

SUMMARY:
The purpose of the study is to know if there is relation between the dynamics of pelvic floor muscles and different phonation pattern.

DETAILED DESCRIPTION:
Some pelvic floor physical therapists are beginning to experiment with using phonation and vocalization cues to elicit different pelvic floor movements . However, there is a significant gap in the literature about the coordination and movement between the pelvic floor and glottis during speech and phonation, and there is an urgent need to identify the voices accompanied by increasing pelvic floor tone and integrating them into pelvic floor strengthening programs and voices accompanied by lowering pelvic floor tone and integrating them into pelvic floor down-training programs. To date, there has been only one study describing pelvic floor displacement during vocalization tasks. So this study aims to investigate pelvic floor muscle displacement during respiratory and phonatory tasks using trans-abdominal ultrasound to assess respiratory and phonatory tasks that can relax or enhance pelvic floor tone and be integrated into clinical practice.

ELIGIBILITY:
Inclusion Criteria:

- 1. They should be virgin, healthy female physiotherapy students. 2. They have regular menstruation (3-8 days in duration, with 21-35 days in-between).

3. Their ages will range from 18 to 25 years old. 4. Their body mass index (BMI) will range from 18 to 24.9 Kg/m2. 5. Their waist- hip ratio will be less than (0.8).

Exclusion Criteria:

1. Any urological, gynecological, respiratory, or vocal disorders in the previous 12 weeks.
2. Pelvic floor dysfunction.
3. Professionally trained singers.

   -

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Twenty healthy female university students will participate in this study. They will be selected from faculty of physical therapy, Cairo University.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-12-03 (Estimated); Primary Completion 2025-01-03 (Estimated); Study Completion 2025-01-10 (Estimated)

PRIMARY OUTCOMES:
Assessment of pelvic floor muscle displacement | 1 month
  Pelvic floor displacement during phonation will be assessed using trans-abdominal ultrasound with a 3.5-MHz transducer. Posterior bladder wall displacement will be measured in the sagittal plane with standardized markers at rest and maximal distortion. A bladder filling protocol will ensure imaging clarity. Participants will perform pelvic floor tasks (e.g., contraction, strain, Valsalva) and phonation/respiratory exercises (e.g., "ah" sounds, coughing, SOVT exercises). Tasks will last 3 seconds, be repeated thrice, and baseline and end measurements will be recorded.

SECONDARY OUTCOMES:
Voice pitch classification | 1 month
  the females' voice pitch will be classified by having them read "The North Wind and the Sun" three times consecutively in a quiet room, using a Samsung Note 20 mobile phone application for recording. The microphone is placed 30 centimeters from their mouths. The application measures average, median, highest (95th percentile), and lowest (95th percentile) frequencies in Hz to provide a comprehensive analysis of voice pitch and volume, aiding in assessing voice quality and potential disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Doaa A Osman, PhD, Study Director — Ass. prof.; Amel M Yousef, PhD, Study Chair — professor
Locations (1):
- Faculty of physical therapy Cairo university, Giza, Egypt